CLINICAL TRIAL: NCT07185997
Title: A Global, Phase 3, Randomized, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Firmonertinib Compared With Investigator's Choice of Osimertinib or Afatinib as First-Line Treatment in Participants Who Have Locally Advanced or Metastatic Non-Small-Cell Lung Cancer With Epidermal Growth Factor Receptor P-Loop and Alpha C-Helix Compressing (PACC) Uncommon Mutations (ALPACCA)
Brief Title: Study to Evaluate Efficacy and Safety of Firmonertinib Compared With Investigator's Choice of EGFR Inhibitor as First-Line Treatment in Participants Who Have Locally Advanced or Metastatic NSCLC With EGFR P-Loop and Alpha C-Helix Compressing (PACC) Uncommon Mutations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ArriVent BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FURMO-006
Record Dates: First submitted 2025-08-15; First posted 2025-09-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Non-Small-Cell Lung Cancer; Metastatic Non-Small-Cell Lung Cancer; Advanced Non-Small-Cell Lung Cancer; EGFR P-Loop and Alpha C-Helix Compressing; EGFR PACC; EGFR Uncommon Mutations
Keywords: Non-Small Cell Lung Cancer (NSCLC); PACC; Firmonertinib; Furmonertinib; AST2818; FURMO-006; Drug-Therapy; Metastatic Non-Small Cell Lung Cancer; Advanced Non-Small Cell Lung Cancer; NSCLC; Osimertinib; Afatinib; metastatic NSCLC first-line treatment; Carcinoma NSCLC; Respiratory tract neoplasms; Bronchial Neoplasms; Protein Kinase Inhibitors; tyrosine kinase inhibitor (TKI); Alflutinib; Lung neoplasms; EGFR; EGFR kinase domain mutations; EGFR activating mutation; EGFR mutation of unknown significance; Non-classical EGFR mutation; EGFR uncommon mutations; EGFR atypical mutations; G719X; S768I; E709X; E709_T710delinsD; G779F; L747X; V774M; L747P/S; R776C/H; G724S; E736K; I740_K745dup; N771G; K757M/R; V769L/M
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Bronchial Neoplasms; Lung Neoplasms | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Firmonertinib 240 mg (Experimental)
  Interventions: Drug: Firmonertinib
- EGFR-TKI inhibitor osimertinib or afatinib based on investigator's choice (Active Comparator)
  Interventions: Drug: EGFR-TKI inhibitor based on investigator's choice

INTERVENTIONS:
Drug: Firmonertinib — 240 mg oral, daily firmonertinib tablet
  Other Names: AST2818
  Arms: Firmonertinib 240 mg
Drug: EGFR-TKI inhibitor based on investigator's choice — osimertinib 80 mg oral, daily tablet OR afatinib 40 mg oral, daily tablet
  Arms: EGFR-TKI inhibitor osimertinib or afatinib based on investigator's choice

SUMMARY:
Global, Phase 3, randomized, multicenter, open-label study evaluating the efficacy and safety of firmonertinib at a dose level of 240 mg QD compared to investigator's choice of osimertinib (80 mg QD) or afatinib (40 mg QD) in participants who have locally advanced or metastatic NSCLC with EGFR PACC mutations, and who have not received any prior therapy for advanced disease. Participants will be randomized in a 1:1 ratio to treatment with firmonertinib or osimertinib or afatinib and will take the assigned dose daily.

ELIGIBILITY:
Key Eligibility Criteria:

* Histologically or cytologically documented, locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy.
* Documented results of the presence of an Epidermal Growth Factor Receptor (EGFR) PACC mutation in tumor tissue or blood from local testing.
* No prior systemic anticancer therapy regimens received for locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) including prior treatment with any Epidermal Growth Factor Receptor (EGFR)-targeting agents (e.g., previous (EGFR) TKIs, monoclonal antibodies, or bispecific antibodies).
* Patients who have received prior neo-adjuvant and/or adjuvant chemotherapy, immunotherapy, or chemo radiotherapy for non-metastatic disease must have experienced a treatment free interval of at least 12 months.
* Patients with asymptomatic CNS metastases are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) determined by blinded independent central review (BICR) | Until progression or death, assessed up to approximately 4 years
  PFS is defined as the time from randomization to the first occurrence of disease progression as determined by BICR using RECIST v1.1, or death from any cause, whichever occurs first.
Confirmed overall response rate (ORR) as determined by BICR | Until progression or death, assessed up to approximately 3 years
  Confirmed ORR is defined as the percentage of participants with a confirmed CR or PR based on BICR assessment relative to the total number of participants.

SECONDARY OUTCOMES:
Overall survival (OS) | Until death, assessed up to approximately 5 years
  OS is defined as the time from randomization to death from any cause.
Investigator-assessed PFS | Until progression or death, assessed up to approximately 4 years
  Investigator-assessed PFS is defined as the time from randomization to the first documented disease progression or death, whichever occurs first, based on investigator assessment per RECIST v1.1.
Investigator-assessed confirmed ORR | Until progression or death, assessed up to approximately 3 years
  Investigator-assessed confirmed ORR is defined as the percentage of participants with a confirmed CR or PR based on investigator assessment relative to the total number of participants.
Duration of response (DOR) | Until progression or death, assessed up to approximately 4 years
  DOR is defined as the time from first documented evidence of CR or PR until the first documented evidence of disease progression or death, whichever occurs first.
Time to second Progression-free survival (PFS2) | Assessed up to approximately 5 years
  PFS2 is defined as the time from randomization to second progression (ie, earliest of the subsequent progression events after initiation of a new anti-cancer treatment), or death from any cause, whichever occurs first.
Incidence and severity of adverse events (AEs), as a measure of safety and tolerability of firmonertinib | Assessed up to approximately 5 years
  An AE is defined as any unfavorable or unintended medical occurrence in a trial participant administered a pharmaceutical product, regardless of causal attribution.
Change from baseline in safety-related clinical laboratory test results | Assessed up to approximately 5 years
  Safety-related laboratory parameters include absolute neutrophil count, hemoglobin, platelet count, albumin, blood urea nitrogen (BUN), chloride, creatinine, potassium, sodium, alkaline phosphatase (ALP), alanine aminotransferase (ALT); aspartate aminotransferase (AST), total bilirubin. Each parameter is measured using its standard unit. Changes in participants' laboratory test values are evaluated by comparing baseline (pre-treatment) results with those obtained at prespecified time points during or following the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Lam, Study Director — ArriVent BioPharm
Locations (23):
- United States (8):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Texas Oncology, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
- Humanity and Health Clinical Trial Centre, Central, Hong Kong
- Japan (7):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Kurume University Hospital, Kurume-Shi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Tokyo Metropolitan Komagome Hospital, Bunkyō-Ku, Tokyo
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Curie Oncology (Farrer), Singapore
- South Korea (2):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Gachon University Gil Medical Center, Incheon
- Hospital Universitario y Politecnico La Fe, Valencia, Spain
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan
- University College London Hospitals NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided